CLINICAL TRIAL: NCT04901221
Title: Dentoalveolar and Skeletal Changes Associated With a Statically Determinate Force System in the Closure of Anterior Open Bite in Adults: A Single-arm Clinical Trial
Brief Title: The Use of Statically Determinate Force System in Closure of Anterior Open Bite in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Tasnim Yousry, Demonstrator of orthodontics, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Extrusionarchadults
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Anterior Openbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extrusion arch (Experimental): Hand made stainless steel extrusion arch wire (0.016x0.22")
  Interventions: Device: Extrusion arch

INTERVENTIONS:
Device: Extrusion arch — one couple force system is applied; a custom-made extrusion wire from 0.016x0.022 stainless steel wire with helical bends placed 2-5 mm mesial to the molar tube placed in the upper and lower arches and tied distal to the lateral incisors

SUMMARY:
The aim of the current study was to evaluate and quantify the cephalometric changes produced by maxillary and mandibular extrusion arches in closure of anterior open bite in non-growing patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with anterior open bites more than 1 mm, permanent dentition except for the third molars which were extracted if erupted

Exclusion Criteria:

* Frankfort to mandibular plane angle > 40
* congenital craniofacial malformations or temporomandibular joint disorders,
* patients with severe gum show during smiling or increased incisal show at rest.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
angular and vertical linear effects on incisors | up to 6 months
  Extrusion of upper and lower incisors measured from: incisal edge, centroid point and apex to the palatal and mandibular planes for the upper and lower incisors respectively. Angles between long axis of upper incisor to SN plane and palatal plane, Angle between long axis of lower incisor and mandibular plane using lateral cephalometric xray
angular and vertical linear effects on first molars | up to 6 months
  For the first molars: Angular measurements between the long axis of the measuring jigs and the palatal plane and mandibular plane for the upper and lower molars, respectively. Vertical measurements: perpendicular vertical distance from the measuring jigs to the palatal and mandibular planes for the upper and lower molars, respectively, using lateral cephalometric xray.

SECONDARY OUTCOMES:
change in the SN' to Mandibular plane angle | up to 6 months
  measuring the change in the angle between SN' to Mandibular plane angle, using lateral cephalometric xray
change in the palatal to Mandibular plane angle | up to 6 months
  measuring the change in the angle between the palatal to Mandibular plane angle, using lateral cephalometric xray
change in the Anterior facial height | up to 6 months
  measuring the change in the vertical distance between Nasion and Menton, using lateral cephalometric x-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Y Hammad, BDS, Principal Investigator — Alexandria University; Hanan Ismail, PHD, Study Director — Alexandria University; Wessam Marzouk, PHD, Study Chair — Alexandria University; Hassan Moussa, PHD, Study Chair — Alexandria University
Locations (1):
- Alexandria faculty of Dentistry, Alexandria, Egypt